CLINICAL TRIAL: NCT04004923
Title: Monopolar or Bipolar Hysteroscopy: Comparison of the Impact of Two Methods on Intracranial Pressure
Brief Title: Intracranial Pressure in Monopolar and Bipolar Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Huseyin Kiyak, Principal Investigator, M.D., Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Huseyin4
Record Dates: First submitted 2019-06-30; First posted 2019-07-02 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Intracranial Pressure Increase
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monopolar hysteroscopy (Active Comparator): This group of patients will receive Monopolar hysteroscopy for uterine distention.
  Interventions: Procedure: Monopolar hysteroscopy
- Bipolar hysteroscopy (Active Comparator): This group of patients will receive Monopolar hysteroscopy for uterine distention.
  Interventions: Procedure: Bipolar hysteroscopy

INTERVENTIONS:
Procedure: Monopolar hysteroscopy — Unipolar resectoscopes are used in this group and the distention fluid is mannitol
  Arms: Monopolar hysteroscopy
Procedure: Bipolar hysteroscopy — Bipolar resectoscopes are used in this group and the distention fluid is serum physiologic
  Arms: Bipolar hysteroscopy

SUMMARY:
Two distinction fluids are used in operative hysteroscopy. One is monopolar and the second is bipolar. The monopolar fluid contains mannitol and the bipolar fluid contains serum physiologic. This study aims to compare intracranial pressure in patients undergoing monopolar and bipolar hysteroscopy.

DETAILED DESCRIPTION:
Operative hysteroscopy is currently used in the treatment of several diseases including submucosal myomas, polyps, uterine septum, and abnormal intrauterine bleeding. Two different methods for distension of the uterus for hysteroscopy are available currently. One is monopolar and the second is bipolar. The monopolar fluid contains mannitol and the bipolar fluid contains serum physiologic. Passage of the distention fluid into the uterine veins during hysteroscopy might lead to volume overload, water intoxication, hyponatremia, pulmonary edema or brain edema. However, the effect of monopolar hysteroscopy or bipolar hysteroscopy on intracranial pressure in patients undergoing hysteroscopy is unknown. Optic nerve sheath diameter (ONSD) measurement is a surrogate marker of invasive intracranial pressure. This study aims to compare the impact of monopolar and bipolar hysteroscopy on intracranial pressure by using ONSD measurement in patients undergoing hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled to hysteroscopy for treatment of uterine myoma, polyp, septum, or for endometrial ablation.

Exclusion Criteria:

* Postmenopause;
* Kidney disease;
* Cardiovascular disease;
* Glaucoma

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Intracranial pressure | ONSD will be measured 3 times in the two groups. Before completion of hysteroscopy, 2 hours after hysteroscopy and 6 hours after hysteroscopy
  The difference in intracranial pressure between the two study arms measured with optic nerve sheath diameter (ONSD). ONSD is measured using a linear ultrasound probe and reflects intracranial pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Kiyak, MD, Principal Investigator — Kanuni Sultan Suleyman Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No